CLINICAL TRIAL: NCT05182229
Title: Comparing Two Ways to Manage Lymphedema in Head and Neck Cancer Survivors
Brief Title: Comparing Two Ways to Manage Head and Neck Lymphedema
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Jie Deng, Associate Professor, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 20321
Record Dates: First submitted 2021-12-12; First posted 2022-01-10 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Head and Neck Cancer; Lymphedema
MeSH Terms: conditions — Head and Neck Neoplasms; Lymphedema | interventions — carbohydrate-deficient transferrin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Clinic-Based Lymphedema Therapy (Active Comparator)
  Interventions: Other: Clinic-based CDT
- Home-Based (a hybrid model) Lymphedema Therapy (Active Comparator)
  Interventions: Other: Home-based (a hybrid model) CDT

INTERVENTIONS:
Other: Home-based (a hybrid model) CDT — Participants will be provided therapist-administered, in person complete decongestive therapy (CDT) two times per week for two weeks (4 sessions), followed by real-time, virtual CDT consultations two times per week for three weeks (7 sessions) and one in person follow-up visit.
  Arms: Home-Based (a hybrid model) Lymphedema Therapy
Other: Clinic-based CDT — Participants will be provided therapist administered, in-person CDT two times per week for six weeks (12 sessions).
  Arms: Clinic-Based Lymphedema Therapy

SUMMARY:
This randomized clinical trial aims to compare clinic-based CDT and home-based (a hybrid model) CDT on changes in the severity of lymphedema, symptom burden, functional status, and healthcare utilization in HNC survivors with lymphedema.

DETAILED DESCRIPTION:
Primary aim: To compare the effects of clinic-based and home-based (a hybrid model) CDT on changes in the severity of lymphedema.

Secondary aim: To compare the effects of clinic-based and home-based (a hybrid model) CDT on symptom burden and functional status.

Exploratory aim: To compare the healthcare utilization between patients receiving clinic-based versus home-based (a hybrid model) CDT

ELIGIBILITY:
Inclusion Criteria:

* >18 years of age
* <=24 months post-HNC treatment
* Diagnosis of head and neck lymphedema and referral by their oncology providers
* Able to perform self-manual lymphatic drainage
* Having an electronic device (a computer, tablet, iPad, laptop, or smartphone) and internet access at home

Exclusion Criteria:

* Active infection in soft tissues in the head and neck region
* History of moderate or severe carotid artery occlusion
* Significantly severe lymphedema (e.g., severe periorbital swelling)
* Conditions impacting the safe delivery of lymphedema therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2022-03-11 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Changes in severity of lymphedema | Baseline, Immediately after End of Intervention (an average of 6 weeks), 6-Month Post-Intervention, 12-Month Post-Intervention
  Compare the effects of clinic-based and home-based CDT on changes in the severity of lymphedema. This outcome measure will be assessed via Head and Neck - External Lymphedema and Fibrosis Assessment Criteria (HN-LEF Assessment Criteria).

SECONDARY OUTCOMES:
Changes in severity of symptom burden | Baseline, Immediately after End of Intervention (an average of 6 weeks), 6-Month Post-Intervention, 12-Month Post-Intervention
  Compare the effects of clinic-based and home-based CDT on changes in the severity of symptom burden. This outcome measure will be assessed via Head and Neck - Lymphedema and Fibrosis Symptom Inventory (HN-LEF Symptom Inventory)
Changes in degrees of jaw range of motion | Baseline, Immediately after End of Intervention (an average of 6 weeks), 6-Month Post-Intervention, 12-Month Post-Intervention
  Compare the effects of clinic-based and home-based CDT on jaw range of motion. Jaw range of motion will be measured via Jaw Range of Motion Scale.
Changes in degrees of cervical range of motion | Baseline, Immediately after End of Intervention (an average of 6 weeks), 6-Month Post-Intervention, 12-Month Post-Intervention
  Compare the effects of clinic-based and home-based CDT on cervical range of motion. Cervical Range of Motion will be measured via Cervical Range of Motion Instrument.

OTHER OUTCOMES:
Healthcare utilization | Baseline, Immediately after End of Intervention (an average of 6 weeks), 6-Month Post-Intervention, 12-Month Post-Intervention
  Compare healthcare utilization between patients receiving clinic-based versus home-based CDT. Healthcare Utilization Questionnaire will be used in this study.
Healthcare utilization | Baseline, Immediately after End of Intervention (an average of 6 weeks), 6-Month Post-Intervention, 12-Month Post-Intervention
  Compare healthcare utilization between patients receiving clinic-based versus home-based CDT. Electronic Health Records (EHR) will be used in this study.

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Jefferson Cherry Hospital Jefferson Health, Cherry Hill, New Jersey
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Jefferson Health, Philadelphia, Pennsylvania
  - Jefferson Torresdale Hospital Jefferson Health, Philadelphia, Pennsylvania
  - Temple University Hospital and Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Asplundh Cancer Pavilion Jefferson Health, Willow Grove, Pennsylvania

IPD SHARING:
Plan to Share IPD: Undecided